CLINICAL TRIAL: NCT02578784
Title: Prospective, Randomized Trial on the Clinical Utility of Drug-coated Balloons After Angioplasty of Plain Old Balloon-resistent Dialysis Fistula Stenosis Using Cutting Ballons
Brief Title: DEB-after-Cutting Balloon-PTA in Dialysis Fistula Stenosis
Acronym: DEB-after-CB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Claas Philip Nähle, Attending, Department of Radiology and Nuclear Medicine, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKSG 15/086
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Renal Insufficiency
Keywords: Dialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- POBA-after-Cutting Balloon (Placebo Comparator): After cutting balloon angioplasty, subsequent angioplasty is performed using a standard, non-coated balloon (plain old balloon, POBA).
  Interventions: Device: Angioplasty with plain old balloon
- DCB-after-Cutting Balloon (Active Comparator): After cutting balloon angioplasty, subsequent angioplasty is performed using a drug-coated balloon (DCB)
  Interventions: Device: Angioplasty with drug-coated balloon

INTERVENTIONS:
Device: Angioplasty with drug-coated balloon — Angioplasty with drug-coated balloon "Elutax" (Aachen Resonance, Germany)
  Other Names: drug-coated balloon "Elutax"
  Arms: DCB-after-Cutting Balloon
Device: Angioplasty with plain old balloon — Angioplasty with plain old balloon "Sterling" (BostonScientific, Switzerland)
  Other Names: balloon "Sterling"
  Arms: POBA-after-Cutting Balloon

SUMMARY:
The incidence of hemodynamically relevant dialysis fistula stenoses/obstructions after 1 year is between 60-90% (from 62.5 to 91% radiocephalic, brachiocephalic 70-84%, PTFE shunts 62-87%), necessitating a therapeutic measure to preserve dialysis access during this period in 1/3 of the patients. This therapeutic measure is a dilatation of the stenosis using a standard PTA balloon (POBA, plain old balloon angioplasty with a primary technical success rate of 50-79% [2-4].In turn, in 21-50% of the cases an insufficient PTA result is obtained (so-called POBA-resistant stenosis). In these cases, predilatation with a so-called cutting balloon (carrying with small knives on its surface) is performed, leading to a success rate of 89%. However, a problem is the high incidence of restenosis, which is about 40% for recurrent stenosis and over 10% in de novo stenosis.

The use of drug-coated balloon (DCB) in non-POBA resistant stenoses lead to a reduction in the restenosis rate of 35% to 5%. However, the effect of DCB in POBA resistant stenoses is unknown.

Therefore, the aim of this study is to evaluate the clinical benefit of the combined use of a cutting balloon and a drug-coated balloon in POBA resistant dialysis fistula stenoses compared to the sole use of a cutting balloon.

ELIGIBILITY:
Inclusion Criteria:

* dialysis fistula dysfunction requiring cutting balloon angioplasty

Exclusion Criteria:

* missing informed consent or unable to consent
* age < 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Time to worsening of dialysis fistula function [days] | one year

SECONDARY OUTCOMES:
Change in lumen 12 months after PTA [mm] | one year
  aka "late lumen loss"
Change in dialysis flow [ml/min.] | one year
Change in dialysis fistula flow [ml/min.] | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology and Nuclear Medicine, Sankt Gallen, Canton of St. Gallen, Switzerland